CLINICAL TRIAL: NCT02196441
Title: Evaluation of Deep Topical Fornix Nerve Block Versus Topical Anaesthesia in Patients Undergoing Implantable Contact Lens Procedure
Brief Title: Evaluation of Deep Topical Fornix Nerve Block Versus Topical Anaesthesia Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1234656
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Local Anesthesia; Satisfaction
Keywords: deep topical fornix nerve block; topical anesthesia; implantable contact lens procedure
MeSH Terms: conditions — Personal Satisfaction | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Experimental): 0.5% bupivacaine Deep topical fornix nerve block anaesthesia (DTFNB)
  Interventions: Drug: 0.5% bupivacaine
- Group 1 (Experimental): 2% tetracaine local anaesthetic drops
  Interventions: Drug: 2% tetracaine local anaesthetic drops

INTERVENTIONS:
Drug: 2% tetracaine local anaesthetic drops — topical anaesthetic drops
  Other Names: topical anaesthetic drops
  Arms: Group 1
Drug: 0.5% bupivacaine — was performed using two sponges (2x3mm) soaked with 0.5% bupivacaine, applied deep in the conjunctival fornices after anaesthetising the conjunctiva with tetracaine local anaesthetic drops. The sponges were removed after 15 minutes. The anaesthetic effect was tested by grasping the limbus with Castroviejo 0.12 tissue forceps.
  Other Names: Deep topical fornix nerve block anaesthesia
  Arms: Group 2

SUMMARY:
General anaesthesia now a days is not the first choice in phakic intra ocular lens surgery (Phakic IOL) , the short duration of the surgery, general anaesthesia complications, decrease the length of hospital stay and decreasing the costs direct the interest to the regional anaesthesia By the time the traditional retro and peribulbar injections recede to a newer techniques that is safer and cheaper, sub tenon's block using a blunt needle took over due to the more safety profile Even though, still serious problems can occur specially in patients with long axial length.

Deep topical fornix nerve block anaesthesia (DTFNB) and topical anaesthesia gradually took over with promising and successful results, decreasing length of hospital stay and increasing patient satisfaction and fewer margins of complications.

In this study the investigators compared topical anaesthesia alone with DTFNBA in patients undergoing posterior chamber phakic IOL surgery (Visian ICL).

DETAILED DESCRIPTION:
102 patients scheduled for elective ICL/TICL implantation surgery were enrolled in this study after obtaining approval from the institutional ethical committee and written patients consent. the investigators are planning a study of matched sets of patients receiving the case and control treatments with 1 matched control(s) per experimental subject. Prior data indicate that the probability of a treatment failure among controls is 0.05 and the correlation coefficient for exposure between matched experimental and control subjects is 0.1. The true odds ratio for failure in experimental subjects relative to control subjects is 0.1, so the investigators needed to study 51 experimental subjects with 1 matched control(s) per experimental subject to be able to reject the null hypothesis that this odds ratio equals 1 with probability (power) 0.7. The Type I error probability associated with this test of this null hypothesis is 0.3.

All patients were assessed and only those cooperative understanding patients who were deemed suitable for topical and DTFNBA were included in the study. Very anxious patients were omitted from the study.

All the operations were done by one surgeon . Patients were prepared for bilateral implantable contact lens/toric implantable contact lens( ICL/TICL) procedure on the same day.

Group I (1 eye) received topical anaesthetic drops and Group 2 (the second eye) received DTFNBA. Before giving the anaesthetics, a peripheral vein was cannulated and heart rate, oxygen saturation and non-invasive arterial blood pressure were monitored.

Topical anaesthesia was done with 2% tetracaine local anaesthetic drops and DTFNBA was performed using two sponges (2x3mm) soaked with 0.5% bupivacaine, applied deep in the conjunctival fornices after anaesthetising the conjunctiva with tetracaine local anaesthetic drops. The sponges were removed after 15 minutes. The anaesthetic effect was tested by grasping the limbus with Castroviejo 0.12 tissue forceps.

Pain was estimated by the patient using a simple pain score: no pain =0; that does not interfere with the surgical technique, discomfort=1; the surgical technique is performed with difficulty, pain=2; the surgeon is unable to continue the surgical technique . The scoring was done during different stages of surgery: lid retraction while inserting a speculum, tolerance to the microscope light, corneal incision, intraocular lens insertion, tucking of footplates, irrigation aspiration (I/A )of viscoelastic, peripheral iridectomy.

The surgical technique was performed through a clear corneal 3.2 mm tunnel incision, followed by sodium hyalurounate injection, ICL implantation and unfolding, tucking of trailing footplates then side port incision and tucking of leading footplates, myostat injection, then peripheral iridectomy . The total operative time was recorded for every case. If the pain score was 0 or 1, no further management was required but if the pain score was 2 at any stage, 1% preservative free lidocaine was injected intracamerally. Parametric data were analyzed using Students t-test; non parametric data were compared using the Chi-square test. A P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* cooperative understanding patients

Exclusion Criteria:

* Very anxious patients
* coagulopathy
* refusal

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Measure of pain free surgery and Tolerability | during the surgical procedure, 15 minutes
  the patient will be examined for optimum pain free condition (anesthesia)that allow the surgeon to proceed

SECONDARY OUTCOMES:
patient satisfaction | one hour post operative
  Patient satisfaction concerning the procedure using a 2-point scale (1=satisfied, I would want the same anaesthesia/analgesia method for the next surgery, 2=unsatisfied, I would want a different anaesthesia/ analgesia method for the next surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Ali, Lecturer, Principal Investigator — Cairo University
Locations (1):
- Magrabi Aseer ,KSA, Khamis Mushait, West, Saudi Arabia